CLINICAL TRIAL: NCT04100109
Title: Evaluating the Metabolic Effects of Polylactose: A Novel Prebiotic
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution. Study will not be undertaken.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PEDS-2019-27933
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Obesity, Adolescent; Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polylactose (Active Comparator): Subjects randomized to this arm of the study will be asked to consume 15 grams/day of foods containing polylactose
  Interventions: Dietary Supplement: Polylactose
- Placebo (Active Comparator): Subjects randomized to this arm of the study will be asked to consume 15 grams/day of foods containing cellulose, which is an inert dietary fiber, and which will act as our placebo for this project.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Polylactose — Polylactose 15 g/day
  Arms: Polylactose
Other: Placebo — Cellulose 15 g/day
  Arms: Placebo

SUMMARY:
This study will evaluate the feasibility and obtain a preliminary estimate of efficacy of feeding 15 g/day of a new novel prebiotic dietary fiber, termed polylactose, in 40 children (8-12 years old) with obesity (body mass index [BMI]-percentile >/= 95th) who have magnetic resonance imaging (MRI)-confirmed non-alcoholic fatty liver disease [NAFLD] (hepatic fat fraction >/= 5.5%), compared to a placebo of 15 g/d of cellulose, an inert dietary fiber.

DETAILED DESCRIPTION:
Approximately 13% of all children (2 - 19 years old) are afflicted with NAFLD with the prevalence of NAFLD increasing to 60-80% among youth with obesity. NAFLD is characterized by excessive deposition of fat in the liver, which is an independent risk factor for the development of cardiovascular disease (CVD) and type 2 diabetes mellitus (T2DM). Unchecked, NAFLD can progress into more severe forms of liver disease, including NASH, cirrhosis, and hepatocellular carcinoma, which eventually can lead to liver transplantation or death. Unfortunately, treatment of NAFLD through lifestyle interventions is extremely challenging and minimally effective even under intensive conditions. Bariatric surgery has shown promise as a treatment approach in adults, but remains controversial for a treatment of NAFLD in pediatrics.Even if bariatric surgery is proven effective, the overall impact will be low since a very small proportion of adolescents with obesity opt for this extreme treatment. Moreover, surgery is not indicated in youth with milder forms of obesity or younger children and since NAFLD occurs across the entire age-spectrum and is not exclusive to youth with obesity, a large need would be unmet by surgical treatment options. Therefore, novel non-surgical approaches that complement lifestyle modification therapy are needed in order to advance the field in a meaningful way and to provide care to a wide-range of youth with NAFLD. However, no safe or effective pharmacotherapy treatment options are presently available for youth with NAFLD, leaving a tremendous gap in care. Therefore, altering the gut microbiome through administration of a prebiotic dietary fiber is an attractive treatment option.

To date, no medications have been successful at producing meaningful improvements in NAFLD among youth. Similarly, in adults, existing pharmacotherapy options elicit some improvement in liver enzymes and/or histology but have failed to demonstrate widespread efficacy. Moreover, most medications are not indicated for children under the age of 12, and pediatricians are adverse to using them until all other treatment options have failed. Therefore, alternative approaches must be taken in this difficult-to-treat clinical population to identify more effective treatment options. A prebiotic dietary fiber may offer a potential novel treatment option for NAFLD in children with obesity.

Subjects who are interested in participating in the study will be asked to come in for a screening visit where their parent will sign a parental consent form and the child will sign an assent form. Blood will be drawn for safety tests and biomarker sampling. Urine and stool will also be collected. A portable glucose monitor will be placed to collect timed glucose results. Subjects will have an MRI to confirm their NAFLD and their BMI will be calculated. Subjects will undergo a dual x-ray absorptiometry (iDXA) scan and lifestyle counseling. Subjects enrolled in this study will be randomly assigned (1:1) to receive either polylactose or the placebo. Subjects will take the polylactose or the placebo in foods provided by the study team (made in a food-grade space utilizing good manufacturing practices to minimize cross contamination). Subjects will take polylactose/placebo for 26 weeks. They will come have blood drawn for safety tests and biomarkers at weeks 8 and 26. They will have urine and stool samples collected at weeks 8, 20 and 26. Assessments of their glucose levels will be done via a wearable glucose monitor between the screening/randomization and week 4, and again between week 20 and week 26. MRI scans of the liver iDXA scans will be repeated at weeks 8 and 26. Lifestyle counseling and assessment of adverse events, compliance with taking the study product/placebo and tolerability of the intervention will take place at weeks 4, 8, 13, 20 and 26.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-12 years old
* Diagnosis of obesity: BMI percentile >/= 95th (using age- and sex- based Center for Disease Control definitions) or BMI >/= 30 kg/m2
* Elevated alanine aminotransferase (ALT) more than twice the upper limit of normal by gender (>/= 44 U/L for girls, >/= 50 U/L for boys) within 6 months prior to screening or diagnosis of NAFLD from ultrasound or MRI within 6 months of screening or participants with biopsy-proven NASH within 12 months of screening

Exclusion Criteria:

* ALT > 250 U/L at screening
* History of significant alcohol intake or current use
* Impaired fasting glucose (> 100 mg/dL)
* Diabetes (type 1 or 2)
* Current or recent (< 60 months prior to enrollment) use of weight loss medication(s)
* Vitamin E supplementation
* Previous bariatric surgery
* Use of metformin
* Metal or magnetic implants, devices or objects inside of or on the body, which are not MRI compatable
* Recent initiation (< 3 months prior to enrollment) of anti-hypertensive or lipid medication(s)
* Known hypothalamic or pituitary dysfunction
* Tobacco use
* Gilbert's syndrome
* Any known causes of liver disease (except NAFLD and NASH)
* Significant renal dysfunction as calculated by estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73 m2
* Diagnosed monogenic obesity
* History of cancer
* Untreated thyroid disorder
* Current or recent (< 6 months prior to enrollment) use of medication(s) associated with weight gain (e.g. atypical anti-psychotics)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2028-05-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in hepatic fat fraction | Subjects will have MR Spectroscopy at Baseline, Week 8 and Week 26
  The primary efficacy endpoint for this study will be the change in hepatic fat fraction from baseline to week 26

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ryder, PhD, Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: Undecided
The statistical analysis plan and the clinical study report may be shared with other researchers.